CLINICAL TRIAL: NCT07120893
Title: Pilot Study Assessing Acceptability, Feasibility, and Appropriateness of Brief Culturally Adapted Behavioral Activation for Adults With Depression in Primary Care Setting
Brief Title: Pilot Study of Brief Culturally Adapted Behavioral Activation for Adults With Depression in Primary Care Setting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Salma Salma, Principal Investigator, Gadjah Mada University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2396/UN1/PS.1/SD/PT.01.04/2025
Record Dates: First submitted 2025-07-30; First posted 2025-08-13 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Depression in Adults
Keywords: culturally adapted behavioral activation; depressive disorder; primary care; pilot study
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): The intervention arm will receive brief culturally adapted behavioral activation therapy, delivered by primary care psychologist, which consists of three individual face-to-face session. The intervention will include both in session activities and homework activity assignment.
  Interventions: Behavioral: brief culturally adapted behavioral activation

INTERVENTIONS:
Behavioral: brief culturally adapted behavioral activation — The brief culturally adapted behavioral intervention in this study is a three individual-session intervention, delivered in primary health care center by primary care psychologist. Each session will last 30-45 minutes in face-to-face. During each session, participants will learn about behavioral techniques to reduce depression and enhance well-being, and practice it in their daily life through homework activities.

SUMMARY:
This is a pilot study of culturally adapted behavioral activation for adults with depression in primary care setting. As a pilot study following systematic cultural adaptation process, the purpose of this clinical trial is to understand if brief culturally adapted individual intervention based on behavioral activation, can be an acceptable, feasible, and appropriate intervention to reduce depressive symptoms among adults with depression in primary care setting. The main question it aims to answer is:

Is brief culturally adapted behavioral activation intervention delivered by primary care psychologist acceptable, feasible, and appropriate as an evidence based treatment for reducing depressive symptoms among adults with depression in primary care setting?

DETAILED DESCRIPTION:
This is a pilot study using mixed method and single arm design to assess acceptability, feasibility, and appropriateness of brief culturally adapted behavioral activation for adults with depression in primary care setting. In this study, participants will receive three individual sessions of brief culturally adapted behavioral activation intervention delivered by primary care psychologist. The participants and primary care psychologist will be asked to fill standardized questionnaire before and after intervention. In addition, the investigators will ask them after the intervention about their experience in receiving or delivering the intervention using semi-structured interview. The depressive symptom level and quality of life of the participants before and after the intervention will be compared as secondary outcome. The results of this study will serve as reference to revise the intervention manual before testing it in a hybrid effectiveness-implementation trial or the main trial.

ELIGIBILITY:
Inclusion Criteria:

* scored 10 or above on PHQ-9
* provide informed consent

Exclusion Criteria:

* having diagnosed of bipolar disorder, psychotic disorders, or substance abuse disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2025-12-06 (Estimated); Study Completion 2025-12-13 (Estimated)

PRIMARY OUTCOMES:
Participant's and Clinical Provider's Perceived Acceptability as Assessed by Acceptability of Intervention Measure (AIM) | Post-intervention (maximum 1 week after intervention)
  Acceptability is defined as the participant's and clinical provider's perception that a given treatment is agreeable, palatable, or satisfactory and will be measured by Acceptability of Intervention Measure (AIM). AIM consists of four items with five Likert-based responses. The score of the scale will range from 1 to 20 with higher score indicating higher acceptability to the intervention.
Participant's and Clinical Provider's Perceived Feasibility as Assessed by Feasibility of Intervention Measure (FIM) | Post-intervention (maximum 1 week after intervention completed)
  Feasibility is defined as the perceived extent to which the intervention can be successfully used or carried out in primary care setting from participants and clinical providers' perspectives and will be measured by Feasibility of Intervention Measure (FIM). FIM consists of four items with five Likert-type responses. The score of the scale will range from 1 to 20 with higher score indicating higher feasibility of the intervention.
Participant's and Clinical Provider's Perceived Appropriateness as Assessed by Intervention Appropriateness Measure (IAM) | Post-intervention (maximum 1 week after intervention completed)
  Appropriateness is defined as the perceived fit, relevance, or compatibility of brief culturally adapted behavioral activation for adults with depression in primary care setting from participant's and clinical provider's perspectives, and measured by Intervention Appropriateness Measure (IAM). IAM consists of four items with five Likert-based responses. The score of the scale will range from 1 to 20 with higher score indicating higher appropriateness of the intervention.
Qualitative Feedback on Acceptability, Feasibility, and Appropriateness from Participants and Clinical Providers as Assessed using Semi-structured Interview | Post-intervention (maximum 1 week after intervention completed)
  Participants and clinical providers will be asked about their experiences in receiving or providing the intervention through individual qualitative interview to understand their perceived acceptability, feasibility, and appropriateness in a more detailed and comprehensive way.

SECONDARY OUTCOMES:
Change in Depressive Symptoms as Assessed by Patient Health Questionnaire-9 (PHQ-9) | Baseline (week 0) and post-intervention (1 week after intervention completed)
  Participants will fill the PHQ-9 as self-reported questionnaire using paper and pencil format, administered by research assistant. PHQ-9 consists of nine items with four response from 'not at all' (0) to 'nearly every day' (3). The score of the PHQ-9 ranges from 0 to 27 with higher score indicating higher depressive symptoms.
Change in Quality of Life as Assessed by WHO Quality of Life Brief Version (WHOQOL-BREF) | Baseline (week 0) and post-intervention (1 week after intervention completed)
  Participants will fill the WHOQOL-BREV as self-reported questionnaire using paper and pencil format, administered by research assistant. WHOQOL-BREV consists of 26 items with score on each item ranges from 0 to 5. The scale will produce quality of life profile which consists of overall perception of individual's quality of life, overall perception of individual's health, and four quality of life domains (physical health, psychological, social relationship, and environment). The score is calculated using mean score of each domain, then transformed to 4-20. Higher score of the domain indicates higher quality of life.
Change in Anxiety as Assessed by Generalized Anxiety Disorder-7 (GAD-7) | Baseline (week 0) and post-intervention (1 week after intervention completed)
  Anxiety is measured using Generalized Anxiety Disorder-7 (GAD-7) as a self-reported questionnaire using paper and pencil format, administered by research assistant. GAD-7 consists of seven items with four response on each item ranging from 0 to 4. The score of GAD-7 will range from 0 to 21 with higher score indicating higher anxiety.
Change in Depression Diagnosis as Assessed by Structured Clinical Interview for DSM-5 (SCID-5) | Baseline (week 0) and post-intervention (1 week after intervention completed)
  Diagnosis of depression among participants will be compared before and after intervention using SCID-5, administered by primary care psychologist. The result of clinical interview will categorize the participants into active depression or in remission.

OTHER OUTCOMES:
Change in Behavioral Activation as Assessed by Behavioral Activation for Depression Scale - Short Form (BADS-SF) | Every week during the trial from baseline to post-intervention (week 0, 1, 2, 3, and 4)
  The level of behavioral activation among participants will be tracked through the course of treatment using BADS-SF. Participants will fill the BDS-SF every week at the treatment scheduled time. BADS-SF consists of 9 items with response on each item ranging from 0 to 6. The score of the BADS-SF will range from 0 to 54 with higher score indicating higher activation.

CONTACTS AND LOCATIONS:
Locations (1):
- Puskesmas (Primary Healthcare Center), Sleman, Special Region of Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared
Supporting Information: Study Protocol
Time Frame: Beginning at publication date with no end date
Access Criteria: The IPD and supporting information will be shared through Open Science Framework (OSF) Platform.

REFERENCES:
- [Background] Uphoff E, Ekers D, Robertson L, Dawson S, Sanger E, South E, Samaan Z, Richards D, Meader N, Churchill R. Behavioural activation therapy for depression in adults. Cochrane Database Syst Rev. 2020 Jul 6;7(7):CD013305. doi: 10.1002/14651858.CD013305.pub2. PMID 32628293
- [Background] Richards DA, Ekers D, McMillan D, Taylor RS, Byford S, Warren FC, Barrett B, Farrand PA, Gilbody S, Kuyken W, O'Mahen H, Watkins ER, Wright KA, Hollon SD, Reed N, Rhodes S, Fletcher E, Finning K. Cost and Outcome of Behavioural Activation versus Cognitive Behavioural Therapy for Depression (COBRA): a randomised, controlled, non-inferiority trial. Lancet. 2016 Aug 27;388(10047):871-80. doi: 10.1016/S0140-6736(16)31140-0. Epub 2016 Jul 23. PMID 27461440